CLINICAL TRIAL: NCT04294797
Title: Pilotstudie: Presepsin Als möglicher Prädiktor Postoperativer Komplikationen Nach Pankreasresektionen
Brief Title: Presepsin as a Predictor for Postoperative Complications Following Pancreatic Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Presepsin
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Complications
Keywords: Pancreatic resection; POPF; Inflammatory response
MeSH Terms: conditions — Postoperative Complications | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood draw — One additional blood sample for study purpose from the day before surgery, postoperative 1, 3 and 8.

SUMMARY:
The study investigates the local and systemic inflammatory response following pancreatic resections.

DETAILED DESCRIPTION:
Pancreatic resections (PR) are major hepato-pancreatico-biliary (HPB) surgeries associated with significant morbidity and mortality. Despite improvements in surgical technique, as well as peri- and postoperative care, mortality rates range from 2-5%, even in high volume centres. Moreover, morbidity rates after PR can be as high as 70%, especially when evaluated in a prospective setting. In this context, postoperative pancreatic fistula (POPF) represents one of the most frequent complications following PR, with a high variability in the literature ranging from 20% to 64%. Besides POPF, the most frequent complications following PR are delayed gastric emptying (DGE, 18%), postoperative fluid collections (10%), postoperative haemorrhage (PPH, 10%), wound infections (10%), or intra-abdominal abscesses (5%). All of these complications are often characterized by infection and sepsis, and despite all intensive-medical measures, associated with high mortality. In this context, early anticipation and appropriate treatment of clinically relevant grade B or C POPF (CR-POPF) is of utmost importance to prevent fatal outcome.

In order to aid with timely detection and therapy of potentially severe POPF, evaluation of predictive biomarkers that could be able to differentiate early between non-significant biochemical leaks and potentially severe CR-POPF is of urgent interest for all specialties involved in the treatment of pancreatic surgery patients.

Over the last decade, various biomarkers have already been assessed: Procalcitonin (PCT) is one of the most frequently used markers. It has advantages over common infection parameters such as CRP or white blood cells but is often altered in various forms of systemic inflammation and thus not precise enough for an accurate clinical assessment. Connor et al. proposed, that the early postoperative local inflammatory process (postoperative acute pancreatitis, POAP) represents one of the main determinants in POPF development and systemic response measured by CRP could predict severity of POPF. Moreover, in the LEOPARD-2 trial, higher postoperative IL-6 levels were found in patients with severe complications including CR-POPF, whereas IL-8 and CRP Levels in their series were comparable between groups.

More recently, also Presepsin (soluble CD14) showed promising results as a biomarker for sepsis diagnosis and postoperative complications but has never been assessed in the context of major HPB surgeries.

Early detection and therapy of potentially life-threatening complications following major HPB surgery is of urgent interest for all specialties involved in the treatment of these patients and studies investigating the predictive value of Presepsin and other inflammatory markers following PR are lacking. Accordingly, the aim of the present pilot study is to evaluate, for the first time, the kinetics of the biomarker Presepsin after PR and to predict the clinical course.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any pancreatic pathology (benign and malign) requiring surgery
* Written informed consent
* >= 18 years

Exclusion Criteria:

* Pregnancy
* Patients who are not capable of giving informed consent (e.g. with existing medical trustee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Presepsin | Preoperative until postoperative day 8.
  Correlation of Presespin values with postoperative complications, especially POPF.

SECONDARY OUTCOMES:
Biomarker assessment | Preoperative until postoperative day 8.
  Correlation of different biomarkers (CRP, IL-1, IL-6, IL-8, Procalcitonin) with operation associated postoperative complications after pancreatic resections.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gasteiger S, Primavesi F, Gobel G, Braunwarth E, Cardini B, Maglione M, Sopper S, Ofner D, Stattner S. Early Post-Operative Pancreatitis and Systemic Inflammatory Response Assessed by Serum Lipase and IL-6 Predict Pancreatic Fistula. World J Surg. 2020 Dec;44(12):4236-4244. doi: 10.1007/s00268-020-05768-9. Epub 2020 Sep 8. PMID 32901324